CLINICAL TRIAL: NCT07233343
Title: Effect of Fascial Mobilization Therapy on Pain, Grip Strength and Manual Dexterity in Patients With Postpartum Carpal Tunnel Syndrome
Brief Title: Effects of Fascial Mobilization Therapy in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba GÖNEN, Asisst. Prof. Dr., Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/90
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Carpal Tunnel Syndrome (CTS); Fascial Mobilization; Post Partum
Keywords: Carpal Tunnel Syndrome (CTS); fascial mobilization; grip strength; Hand Skills; pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain

STUDY DESIGN:
Intervention Model Description: Participants were divided in two groups. One group will get intervention. One group will be the control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): This group will get conventional physiotherapy that is include range of motion exercises, electrotherapy and resistance exercise training.
  Interventions: Other: Conventional physiotherapy
- Fascial mobilization group (Experimental): This group will get a specific programme that combinated with conventional physiotherapy and fascial mobilization therapy
  Interventions: Other: Fascial mobilization therapy

INTERVENTIONS:
Other: Conventional physiotherapy — Conservative treatment methods such as TENS, normal joint range of motion exercises, tendon gliding exercises and nerve mobilizations will be applied twice a week for 12 weeks, with each session lasting 45 minutes.
  Arms: Control group
Other: Fascial mobilization therapy — In addition to conservative treatment methods, the patients in the study group will receive fascial mobilization techniques, including the flexor retinacula technique, the lacertus fibrosus technique, and 90-120 seconds of application to the epimysial fascia of the wrist flexor muscles. The patients in the study group will receive the same treatment, twice a week for 12 weeks, with each session lasting 45 minutes.
  Arms: Fascial mobilization group

SUMMARY:
The aim of this study, designed as a randomized controlled trial, is to investigate the effects of fascial mobilization treatment on pain, grip strength, and manual dexterity in patients with postpartum carpal tunnel syndrome.

DETAILED DESCRIPTION:
Carpal Tunnel Syndrome (CTS) is a pathological condition characterized by symptoms resulting from compression of the median nerve as it passes through the carpal tunnel. This syndrome is also known as compression neuropathy, the most common type of neuropathy in the upper extremities, and is reported to affect approximately 3% of the adult population. Entrapment neuropathies can affect a specific area of the nerve, but overall, this condition can lead to significant psychological, physical, and financial problems for the patient. The most common etiology of CTS is idiopathic; however, other possible causes include local (tenosynovitis, hypertrophic synovium, etc.), trauma including Colles' fracture, dislocation of the carpal bone(s), recent/malformed fracture near the wrist joint, anatomical anomalies, tumors, and regional and systemic factors. For example, occupational factors such as repetitive stress injuries to the flexor tendons of the hand, such as those seen in computer scientists, data entry clerks, typists, pianists, guitarists, sitarists, and fine art painters, may predispose to the development of CTS. Relevant literature indicates that CTS is three times more common in women than in men. It is known that the risk of CTS is significantly increased in individuals who work in repetitive and strenuous occupations. Furthermore, CTS is considered a common musculoskeletal problem during pregnancy. According to scientific data, the prevalence of CTS in the third trimester of pregnancy is approximately 63%. Approximately 53% of these cases are reported to be unilateral.

Causes of CTS during pregnancy include changes in the musculoskeletal system due to hormonal changes and edema that occur during pregnancy. Additionally, gestational diabetes can contribute to the development of CTS by causing a general slowing of nerve conduction velocity. Symptoms of CTS typically become more severe late in the day and may include pain, numbness, and tingling in the hand. The pain is usually felt along the median nerve path, but it can affect the entire hand and radiate to the arm and shoulder. Symptoms often begin with loss of sensation in the distal fingers. However, in more severe cases, muscle weakness and atrophy of the abductor pollicis brevis muscle, causing loss of palmar abduction of the thumb. CTS in pregnancy has generally been found to be less severe than non-pregnancy-related CTS. A study of both pregnant and non-pregnant women diagnosed with CTS found that pregnant patients recovered approximately 3 to 4 times faster than non-pregnant patients.

The aim of this randomized controlled trial was to investigate the effects of fascial mobilization therapy on pain, grip strength, and dexterity in patients with postpartum carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with CTS by a physician
* Being in the post-pregnancy period (first year)
* Presence of pregnancy-related edema
* Presence of pain, tenderness, and numbness in the median nerve neurodynamic test
* Positive Tinnel and Phalen tests
* Individuals who volunteered to participate in the study

Exclusion Criteria:

* Having a history of CTS before pregnancy
* Being diagnosed with a cervical disc herniation
* Individuals with a history of upper extremity surgery within the last year

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since the study was conducted on patients diagnosed with carpal tunnel in the post-partum period, only female patients were included in the study.
Enrollment: 30 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
The Pain | through of the study, average 12 weeks
  Mc Gill Short Form will used to determine the type and severity of the pain. A short form of the McGill Pain Questionnaire (SF-MPQ) has been developed. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Pain pressure threshold | through of the study, average 12 weeks
  After localizing the painful area by palpation, force will be applied with an algometer until the patient experiences pain and discomfort. The value displayed on the algometer will be recorded, and three measurements will be taken, and the average will be used for analysis. PPT measurement with an algometer is a reliable method for determining tissue nociceptive sensitivity.
Grip strength | through of the study, average 12 weeks
  A Jamar hand dynamometer will be used to measure patients' grip strength. Grip strength is measured with the Jamar hand dynamometer, recommended by the American Association of Hand Therapists (AETD) and whose validity and reliability have been confirmed in numerous studies. This device is considered the gold standard for measuring hand grip strength. Measurements will be taken before and after treatment, and three times, 10 seconds apart. Each measurement will be taken at the same difficulty level. Generally, the average of the three measurements will be taken.
Hand skills | through of the study, average 12 weeks
  The Moberg test has functional value because it reflects manual performance. It relies heavily on motor control of the thumb, index finger, and middle finger. The test is administered in two stages: with eyes open and eyes closed, beginning with the dominant hand. A box, 12 small metal objects (screws, paper clips, key ring, safety pin, small nuts, coins, and a key), and a stopwatch are used to administer the test. Subjects are instructed to pick up each object one by one and place it in the box as quickly as possible without slipping. The time from the initial position until the last object is released is recorded. The test is then repeated with eyes closed. The test is repeated three times, with the best result recorded.
Hand skills | through of the study, average 12 weeks
  The Nine-Hole Peg test, used to assess manual dexterity, involves patients quickly removing nine wooden pegs from a storage box, placing them in random holes, then collecting them from the holes and returning them to the storage compartment. The time is measured in seconds using a stopwatch, and anything over 20 seconds is considered a "loss of skill."

SECONDARY OUTCOMES:
Upper extremity functionality | through of the study, average 12 weeks
  The Questionnaire for Arm, Shoulder, and Hand Disabilities (Q-DASH) will be used to assess individuals' upper extremity functions. This questionnaire is a self-administered measurement tool with validated validity and reliability in Turkish. The validity and reliability of the Turkish version of the DASH questionnaire (DASH-T) was conducted in Turkey by Düger et al. in 2006. The questionnaire, consisting of 30 questions, assesses the individual's ability to perform functional activities (21 items), pain (5 items), and psychosocial aspects of the disease (4 items). The total score ranges from 0 to 100, with a higher score indicating better outcomes.
Carpal tunnel symptom severity | through of the study, average 12 weeks
  Specific to Boston Carpal Tunnel Syndrome (CTS), it consists of two different scales assessing symptom severity and functional capacity. Each item is scored from 1 to 5. The mean score is obtained by dividing the total score by the number of items and ranges from 1 to 5. A high score indicates low functional capacity. Mean scores are calculated separately for symptom severity and functional capacity. The symptom score consists of 11 items, and the function score consists of 8 items.
Wrist edema evaluation | through of the study, average 3 weeks
  A water displacement vessel is used to measure wrist edema. The purpose is to measure and assess extremity volume. This involves filling a container of a predetermined volume with water to the overflow level, then slowly immersing the extremity in the container. The amount of water displaced from the container represents the extremity volume.
Anxiety | through of the study, average 12 weeks
  The Beck Anxiety Inventory is used to measure the anxiety level of patients with postpartum carpal tunnel syndrome. The scale was developed by Aaron Beck. It consists of 21 questions and has international validity. The first validity and reliability study of the scale was conducted by Ulusoy (1993). The answers to the questions in the Beck Anxiety Inventory are scored. "None" is 0 points, "Mild" is 1 point, "Moderate" is 2 points, and "Severe" is 3 points. The scores are totaled at the end of the test. Scores between 8 and 15 are categorized as mild anxiety symptoms, 16-25 as moderate anxiety symptoms, and 26-63 as severe anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba GÖNEN, Asisst. Prof. Dr., Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Branchini M, Lopopolo F, Andreoli E, Loreti I, Marchand AM, Stecco A. Fascial Manipulation(R) for chronic aspecific low back pain: a single blinded randomized controlled trial. F1000Res. 2015 Nov 3;4:1208. doi: 10.12688/f1000research.6890.2. eCollection 2015. PMID 26834998
- [Result] Karjalanen T, Raatikainen S, Jaatinen K, Lusa V. Update on Efficacy of Conservative Treatments for Carpal Tunnel Syndrome. J Clin Med. 2022 Feb 11;11(4):950. doi: 10.3390/jcm11040950. PMID 35207222
- [Result] Abdolrazaghi HA, Khansari M, Mirshahi M, Ahmadi Pishkuhi M. Effectiveness of Tendon and Nerve Gliding Exercises in the Treatment of Patients With Mild Idiopathic Carpal Tunnel Syndrome: A Randomized Controlled Trial. Hand (N Y). 2023 Mar;18(2):222-229. doi: 10.1177/15589447211006857. Epub 2021 Apr 15. PMID 33855879
- [Result] Huisstede BM, Friden J, Coert JH, Hoogvliet P; European HANDGUIDE Group. Carpal tunnel syndrome: hand surgeons, hand therapists, and physical medicine and rehabilitation physicians agree on a multidisciplinary treatment guideline-results from the European HANDGUIDE Study. Arch Phys Med Rehabil. 2014 Dec;95(12):2253-63. doi: 10.1016/j.apmr.2014.06.022. Epub 2014 Aug 12. PMID 25127999
- [Result] Kozak A, Schedlbauer G, Wirth T, Euler U, Westermann C, Nienhaus A. Association between work-related biomechanical risk factors and the occurrence of carpal tunnel syndrome: an overview of systematic reviews and a meta-analysis of current research. BMC Musculoskelet Disord. 2015 Sep 1;16:231. doi: 10.1186/s12891-015-0685-0. PMID 26323649
- [Result] Heebner ML, Roddey TS. The effects of neural mobilization in addition to standard care in persons with carpal tunnel syndrome from a community hospital. J Hand Ther. 2008 Jul-Sep;21(3):229-40; quiz 241. doi: 10.1197/j.jht.2007.12.001. PMID 18652967
- [Result] Ng CL, Ho DD, Chow SP. The Moberg pickup test: results of testing with a standard protocol. J Hand Ther. 1999 Oct-Dec;12(4):309-12. doi: 10.1016/s0894-1130(99)80069-6. PMID 10622197
- [Result] Oxford Grice K, Vogel KA, Le V, Mitchell A, Muniz S, Vollmer MA. Adult norms for a commercially available Nine Hole Peg Test for finger dexterity. Am J Occup Ther. 2003 Sep-Oct;57(5):570-3. doi: 10.5014/ajot.57.5.570. PMID 14527120
- [Result] Yakut Y, Yakut E, Bayar K, Uygur F. Reliability and validity of the Turkish version short-form McGill pain questionnaire in patients with rheumatoid arthritis. Clin Rheumatol. 2007 Jul;26(7):1083-7. doi: 10.1007/s10067-006-0452-6. Epub 2006 Nov 15. PMID 17106618
- [Result] Sheereen FJ, Sarkar B, Sahay P, Shaphe MA, Alghadir AH, Iqbal A, Ali T, Ahmad F. Comparison of Two Manual Therapy Programs, including Tendon Gliding Exercises as a Common Adjunct, While Managing the Participants with Chronic Carpal Tunnel Syndrome. Pain Res Manag. 2022 Jun 8;2022:1975803. doi: 10.1155/2022/1975803. eCollection 2022. PMID 35719196